CLINICAL TRIAL: NCT03818139
Title: Performance of Lung Ultrasonography for Endotracheal Tube Positioning in Neonates
Acronym: ECHOSI
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0022 (ECHOSI)
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Diagnostic Imaging; Newborn; Intubation; Ultrasonography
Keywords: diagnostic imaging, Newborn, Intubation, Ultrasonography methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: radiography thorax — The ultrasound of the thorax will be performed while waiting for the X-ray thorax

SUMMARY:
Lung Ultrasonography (US) has been shown to be effective for verifying endotracheal tube (ETT) position in adults and children but has been less studied in neonates. The aim of this study is to evaluate the performance of lung US in determining correct ETT position in neonates, in comparison with X Ray

ELIGIBILITY:
Inclusion Criteria:

* Newborns
* treated with mechanical ventilation
* and required chest X ray for determining ETT position
* hospitalised in neonatal intensive Care unit , Limoges, France
* signed parental inform consent

Exclusion Criteria:

* Congenital heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborns treated with mechanical ventilation and required chest X ray for determining ETT position
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Concordance of ETT positioning according to lung ultrasonography with chest X ray results | Day 0
  X Ray correct ETT position : ETT's tip will be correctly positioned if located between the upper edge of the first thoracic vertebra and the lower edge of the second thoracic vertebra.
  Ultrasound correct ETT position : ETT'S tip will be correctly positioned if the distance between ETT's tip and the junction of the brachycephalic artery with aortic arch will be measured between 0.8 and 1.5 centimeter

SECONDARY OUTCOMES:
time of realization lung US | Day 0
  time of realization lung US
time of realization chest X ray | Day 0
  time of realization chest X ray
variability inter observator | Day 0
  Concordance of thoracic ultrasound results between the operator and the reviewer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France